CLINICAL TRIAL: NCT00457119
Title: A Two-step Phase 1 Study Investigating the Combination of RAD001 With Carboplatin, Paclitaxel and Bevacizumab in Non-small-cell Lung Cancer (NSCLC) Patients Not Treated Previously With Systemic Therapy
Brief Title: Combination of RAD001 With Carboplatin, Paclitaxel and Bevacizumab in Non-small-cell Lung Cancer (NSCLC) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2114; 2006-002760-26 (EudraCT Number)
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; NSCLC; Advanced Lung Cancer; RAD; RAD001; chemotherapy; carboplatin; paclitaxel; bevacizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Step 1 Arm 1 (Experimental): 5mg/day RAD001 + Carboplatin + Paclitaxel
  Interventions: Drug: RAD001
- Step 1, Arm 2 (Experimental): 30mg/week RAD001 + Carboplatin + Paclitaxel
  Interventions: Drug: RAD001
- Step 2, Arm 1 (Experimental): 5mg/day RAD001 + Carboplatin + Paclitaxel + Bevacizumab
  Interventions: Drug: RAD001
- Step 2, Arm 2 (Experimental): 30mg/week RAD001 + Carboplatin + Paclitaxel + Bevacizumab
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — 5mg oral tablets of RAD001 - for the 5mg/daily arm, 10mg oral tablets x 3 of RAD001 - for the 30mg/weekly arm
  Other Names: Everolimus

SUMMARY:
This 2 step study aims to establish a tolerable dose level and regimen of RAD001 in patients with advanced NCLC not previously treated with systemic therapy. In step 1 of this study, RAD 001 is given in combination with carboplatin and paclitaxel and in Step 2 RAD001 is given in combination with carboplatin, paclitaxel and bevacizumab

DETAILED DESCRIPTION:
This is a two-step, open-label, multi-center, dose escalation Phase 1 study in which RAD001 is administered in combination with carboplatin and paclitaxel (CP) in Step 1 as well as carboplatin, paclitaxel, and bevacizumab (CPB) in Step 2 in patients with advanced (unresectable or metastatic) NSCLC not treated previously with systemic therapy for advanced disease

ELIGIBILITY:
Inclusion criteria:

* Age over 18 years
* Advanced Non Small Cell Lung Cancer (Stage IIIB/IV)
* Ability to perform normal daily functions

Exclusion criteria:

* Chronic steroid treatment
* Prior treatment with chemotherapy for advanced lung cancer
* Prior treatment with mTOR inhibitors
* Active bleeding conditions, skin conditions, gastrointestinal disorders, mouth ulcers, eye conditions, chronic liver or kidney disorders, uncontrolled diabetes, infections or other severe medical conditions
* Known sensitivity to platinum compounds, taxanes or bevacizumab
* Other cancers within the past 5 years
* Pregnant or breastfeeding women Other protocol-defined inclusion/exclusion criteria may apply

Ages: 23 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Establish the feasible doses/regimens of RAD001 in combination with chemotherapy. Primary endpoint is the End-of-cycle DLT rate | Ever 3 months or once a critical DLT occurs

SECONDARY OUTCOMES:
Relative dose intensity (RDI) of Carboplatin + Paclitaxel (step 1) | End of step 1
Relative dose intensity (RDI) of Carboplatin + Paclitaxel + bevacizumab (step 2) | End of Step 2
PK parameters derived from PK profiles of treatment drugs alone and in combination | End of Step 1 and Step 2
Best overall response - measured by CT/MRI scan every 6-8 week | Every 6-8 week

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (4):
  - Georgetown University/Lombardi Cancer Center StudyCoordinator:CRAD001C2114, Washington D.C., District of Columbia
  - LSU HEALTH SCIENCES CENTER/ LSU SCHOOL OF MEDICINE Feist-Weiller Cancer Center, New Orleans, Louisiana
  - U of TX Southwestern Medical Center - SimmonsCompCancerCtr Clinical Research Office, Dallas, Texas
  - MD Anderson Cancer Center/University of Texas Thoractic Head/Neck Med. Onc., Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Heidelberg, Victoria
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg